CLINICAL TRIAL: NCT03041441
Title: Non-invasive Estimation of CSF Pressure Using MRI in Patients With Spontaneous Intracranial Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00078211
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Results first posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Intracranial Hypotension
MeSH Terms: conditions — Intracranial Hypotension | interventions — Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MRICP method (Experimental): MRI sequences have been developed that may be able to estimate ICP in a non-invasive fashion.6-10 The MRI-based method for measurement of ICP (MRICP method) is based on basic principles of the cranio-spinal CSF physiology: The mono-exponential relationship between intracranial volume and pressure leads to a linear relationship between elastance (i.e., the derivative of pressure with respect to volume) and pressure.
  Interventions: Device: MRI algorithm; Procedure: Lumbar puncture; Procedure: Epidural patching

INTERVENTIONS:
Device: MRI algorithm — MRI sequences have been developed that may be able to estimate intracranial pressure in a non-invasive fashion
Procedure: Lumbar puncture — Lumbar puncture according to the standard-of-care treatment plan.
Procedure: Epidural patching — Epidural patching will be performed to the standard-of -care treatment plan

SUMMARY:
The purpose of this study is to estimate the intracranial pressure (ICP, the pressure in your head) in subjects with intracranial hypotension (a condition caused by leakage of the fluid that surrounds your brain and spine) using non-invasive magnetic resonance imaging (MRI) techniques, and to determine whether changes in estimated ICP are seen after treatment of this condition.

DETAILED DESCRIPTION:
Subjects with known intracranial hypotension who are scheduled to undergo standard-of-care CSF pressure measurement using lumbar puncture prior to planned epidural patch treatment will first undergo a research MRI of the brain in order to estimate ICP. The imaging protocol is listed in Appendix 1. All research scans are performed without intravenous contrast. Approximate scan time per session will be 20-22 minutes.

Subjects will then undergo lumbar puncture according to the standard-of-care treatment plan. Estimated values of CSF pressure derived from MRI will be compared to values measured during lumbar puncture. Patients will then undergo standard-of-care epidural patching. A repeat research MRI after epidural patching will be performed to assess for differences in pre- and post-treatment scans.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of intracranial hypotension, established by the following criteria: the presence of orthostatic headache, and one or more of the following criteria: prior CSF opening pressure ≤6 cmH20, demonstration of an active spinal CSF leak on prior spine imaging, or cranial MRI changes of intracranial hypotension.15
* Ability to provide informed consent.
* Expected ability to complete standard-of-care procedures (lumbar puncture and epidural patching)

Exclusion Criteria:

* Known contraindication to MRI (pacemaker, MRI incompatible hardware, etc.)
* Severe claustrophobia or other condition requiring the need for anxiolysis, sedation, or any other medication for MRI scanning
* Inability or expected inability to complete study interventions as scheduled
* Any known contraindication to standard-of-care procedures (e.g. coagulopathy, allergic reaction to required medication, lack of vascular access, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kranz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRICP Method
Started | 5
Completed | 3
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | MRICP Method
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Pressure Measurements Estimated by the MRICP Technique.
Description: The measurement of the momentary differences between the volumes of blood and CSF entering and leaving the cranium during the cardiac cycle provides an estimate of the intracranial volume change, and the pressure difference is estimated using the derivative of the CSF velocities.
Time Frame: During scan, approximately 30 minutes
Population: Data not collected on 4 participants.
Measure: Number; unit: cm H20
Arm/Group | MRICP Method
Number analyzed (Participants) | 1
cm H20 | 6.5

2. Primary Outcome: Cerebro Spinal Fluid Pressure Measured by Lumbar Puncture
Description: The CSF pressure measured at lumbar puncture (LP), is 100-180 mm of H2O (8-15 mm Hg) with the patient lying on the side and 200-300 mm with the patient sitting up.
Time Frame: During lumbar procedure, up to 2 hours
Population: Data not collected on 4 participants.
Measure: Number; unit: cm H20
Arm/Group | MRICP Method
Number analyzed (Participants) | 1
cm H20 | 19.0

3. Secondary Outcome: Change in Intracranial Pressure Estimated With MR Technique
Description: Description: assessment of change in estimated ICP prior to and following standard-of-care epidural patching; and (2) evaluate changes in diameter and flow velocity through the transverse dural venous sinus prior to and following epidural blood patching.
Time Frame: Baseline, 24 hours
Population: Data not collected.
Arm/Group | MRICP Method
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Caliber to the Transverse Venous Sinus Caliber
Description: Change in caliber to the Transverse Venous Sinus caliber has measured by non-contrast 3D phase contrast MR venography.
Time Frame: Baseline, 24 hours
Population: Data not collected on 2 participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MRICP Method
Number analyzed (Participants) | 3
mm | 1.1 (0.5)

5. Secondary Outcome: Change in Flow Velocity Through the Transverse Dural Venous Sinus
Description: Description:Change in Flow velocity through the Transverse Dural venous sinus has measured by non-contrast 3D phase contrast MR venography
Time Frame: Baseline, 24 hours
Population: Data not collected.
Arm/Group | MRICP Method
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 30 hours
Arm/Group | MRICP Method
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT03041441/Prot_000.pdf